CLINICAL TRIAL: NCT03334851
Title: A PHASE 1, RANDOMIZED, MULTI-CENTER, DOUBLE-BLIND, SPONSOR OPEN, PLACEBO-CONTROLLED, SINGLE AND MULTIPLE DOSE-ESCALATION STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS AND PHARMACODYNAMICS OF PF-06835375 IN SUBJECTS WITH SEROPOSITIVE SYSTEMIC LUPUS ERYTHEMATOSUS OR RHEUMATOID ARTHRITIS
Brief Title: Safety and Tolerability Study Of PF-06835375 In Subjects With Seropositive Systemic Lupus Erythematosus Or Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: C1131001; 2017-003077-34 (EudraCT Number)
Record Dates: First submitted 2017-11-03; First posted 2017-11-07 (Actual); Results first posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-01

CONDITIONS: Systemic Lupus Erythematosus; Rheumatoid Arthritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Part A, Cohort 1 (Experimental): Subjects will receive a single dose of PF-06835375 or placebo on Day 1 via intravenous administration
  Interventions: Drug: PF-06835375; Drug: Placebo
- Part A, Cohort 2 (Experimental): Subjects will receive a single dose of PF-06835375 or placebo on Day 1 via intravenous administration.
  Interventions: Drug: PF-06835375; Drug: Placebo
- Part A, Cohort 3 (Experimental): Subjects will receive a single dose of PF-06835375 or placebo on Day 1 via intravenous administration.
  Interventions: Drug: PF-06835375; Drug: Placebo
- Part A, Cohort 4 (Experimental): Subjects will receive a single dose of PF-06835375 or placebo on Day 1 via intravenous administration.
  Interventions: Drug: PF-06835375; Drug: Placebo
- Part A, Cohort 5 (Experimental): Subjects will receive a single dose of PF-06835375 or placebo on Day 1 via intravenous administration.
  Interventions: Drug: PF-06835375; Drug: Placebo
- Part A, Cohort 6 (Experimental): Subjects will receive a single dose of PF-06835375 or placebo on Day 1 via intravenous administration.
  Interventions: Drug: PF-06835375; Drug: Placebo
- Part A, Cohort 7 (Experimental): Subjects will receive a single dose of PF-06835375 or placebo on Day 1 via intravenous administration.
  Interventions: Drug: PF-06835375; Drug: Placebo
- Part A, Cohort 8 (Experimental): Subjects will receive a single dose of PF-06835375 or placebo on Day 1 via intravenous administration.
  Interventions: Drug: PF-06835375; Drug: Placebo
- Part B, Cohort 1 (Experimental): Subjects will receive two doses of PF-06835375 or placebo on Day 1 and Day 29 via subcutaneous administration.
  Interventions: Drug: PF-06835375; Drug: Placebo
- Part B, Cohort 2 (Experimental): Subjects will receive two doses of PF-06835375 or placebo on Day 1 and Day 29 via subcutaneous or intravenous administration.
  Interventions: Drug: PF-06835375; Drug: Placebo
- Part B, Cohort 3 (Experimental): Subjects will receive two doses of PF-06835375 or placebo on Day 1 and Day 29 via subcutaneous or intravenous administration.
  Interventions: Drug: PF-06835375; Drug: Placebo
- Part B, Cohort 4 (Experimental): Subjects will receive two doses of PF-06835375 or placebo on Day 1 and Day 29 via subcutaneous or intravenous administration.
  Interventions: Drug: PF-06835375; Drug: Placebo
- Part B, Cohort 5 (Experimental): Subjects will receive two doses of PF-06835375 or placebo on Day 1 and Day 29 via subcutaneous or intravenous administration.
  Interventions: Drug: PF-06835375; Drug: Placebo
- Part B, cohort 6 (Experimental): Subjects will receive two doses of PF-06835375 or placebo on Day 1 and Day 29 via subcutaneous or intravenous administration.
  Interventions: Drug: PF-06835375; Drug: Placebo

INTERVENTIONS:
Drug: PF-06835375 — Intravenous (IV) or subcutaneous (SC) administration. Subjects will receive one or two doses. Doses will be ascending and determined by emerging data.
Drug: Placebo — Matching placebo for PF-06835375 IV or SC. Subjects will receive one or two doses.

SUMMARY:
This is a Phase 1 single and multiple dose escalation study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of PF-06835375 in subjects with seropositive SLE or RA. The design is double-blind, sponsor open and placebo controlled. This study will include two parts: Part A and Part B. Part A will consist of single ascending dose cohorts, Part B of multiple ascending dose cohorts. This study will enroll up to a total of approximately 112 subjects at approximately 10 sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Rheumatoid Arthritis: confirmed diagnosis according to 2010 ACR/EULAR criteria with symptom duration at least 6 months and positive with Rheumatoid Factor and/or anti citrullinated peptide antibody
* Patients with Systemic Lupus Erythematosus: Confirmed diagnosis according to the SLICC Classification Criteria with symptom duration at least 6 months and at least one of the following: positive antinuclear antibody titer, positive anti-dsDNA, anti-Smith antibodies

Exclusion Criteria:

* Active central nervous system manifestations, systemic vasculitis or pleuro/pericarditis
* Active lupus nephritis
* Treatment with B cell depleting agents within 52 weeks prior to screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-11-17 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- United States (16):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Wallace Rheumatic Studies Center, Beverly Hills, California
  - Prive aftercare, Los Angeles, California
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Private Practice of Robert W. Levin, MD, Clearwater, Florida
  - Avail Clinical Research, DeLand, Florida
  - Omega Research Maitland, LLC, Orlando, Florida
  - Larkin Hospital, South Miami, Florida
  - Qps Mra, Llc, South Miami, Florida
  - Qps-Mra, Llc, South Miami, Florida
  - PAREXEL International - EPCU Baltimore, Baltimore, Maryland
  - Rheumatology Express, Catonsville, Maryland
  - Carolina Phase 1 Research, LLC, Raleigh, North Carolina
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas
  - MPP Infusion Centers, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Cohen S, Beebe JS, Chindalore V, Guan S, Hassan-Zahraee M, Saxena M, Xi L, Hyde C, Koride S, Levin R, Lubaczewski S, Salganik M, Sloan A, Stevens E, Peeva E, Vincent MS, Martin DA, Chu M. A Phase 1, randomized, double-blind, placebo-controlled, single- and multiple-dose escalation study to evaluate the safety and pharmacokinetics/pharmacodynamics of PF-06835375, a C-X-C chemokine receptor type 5 directed antibody, in patients with systemic lupus erythematosus or rheumatoid arthritis. Arthritis Res Ther. 2024 Jun 6;26(1):117. doi: 10.1186/s13075-024-03337-2. PMID 38845046
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C1131001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included two parts: Part A, consisting of 7 single ascending dose (SAD) cohorts (placebo and PF-06835375 0.03 mg, 0.1 mg, 0.3 mg, 1 mg, 3 mg, 6 mg); and Part B, consisting 6 multiple ascending dose (MAD) cohorts (placebo and PF-06835375 0.3 mg, 1 mg, 3 mg, 6 mg, 10 mg). In Part A (SAD), 32 participants were assigned to treatment, 1 of whom was not treated. In Part B (MAD), 42 participants were screened and treated.
Groups:
- Placebo IV SAD: Participants received single dose of placebo on Day 1 as an intravenous (IV) infusion.
- PF-06835375 0.03 mg IV SAD: Participants received single dose of PF-06835375 0.03 mg on Day 1 as an IV infusion.
- PF-06835375 0.1 mg IV SAD: Participants received single dose of PF-06835375 0.1 mg on Day 1 as an IV infusion.
- PF-06835375 0.3 mg IV SAD: Participants received single dose of PF-06835375 0.3 mg on Day 1 as an IV infusion.
- PF-06835375 1 mg IV SAD: Participants received single dose of PF-06835375 1 mg on Day 1 as an IV infusion.
- PF-06835375 3 mg IV SAD: Participants received single dose of PF-06835375 3 mg on Day 1 as an IV infusion.
- PF-06835375 6 mg IV SAD: Participants received single dose of PF-06835375 6 mg on Day 1 as an IV infusion.
- Placebo SC MAD: Participants received two doses of placebo subcutaneously (SC) with first dose on Day 1 and the repeated dose on Day 29.
- PF-06835375 0.3 mg SC MAD: Participants received two doses of PF-06835375 0.3 mg SC with first dose on Day 1 and the repeated dose on Day 29.
- PF-06835375 1 mg SC MAD: Participants received two doses of PF-06835375 1 mg SC with first dose on Day 1 and the repeated dose on Day 29.
- PF-06835375 3 mg SC MAD: Participants received two doses of PF-06835375 3 mg SC with first dose on Day 1 and the repeated dose on Day 29.
- PF-06835375 6 mg SC MAD: Participants received two doses of PF-06835375 6 mg SC with first dose on Day 1 and the repeated dose on Day 29.
- PF-06835375 10 mg SC MAD: Participants received two doses of PF-06835375 10 mg SC with first dose on Day 1 and the repeated dose on Day 29.
Period: Overall Study
Arm/Group | Placebo IV SAD | PF-06835375 0.03 mg IV SAD | PF-06835375 0.1 mg IV SAD | PF-06835375 0.3 mg IV SAD | PF-06835375 1 mg IV SAD | PF-06835375 3 mg IV SAD | PF-06835375 6 mg IV SAD | Placebo SC MAD | PF-06835375 0.3 mg SC MAD | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
Started | 8 | 3 | 3 | 3 | 3 | 6 | 5 | 11 | 6 | 6 | 7 | 6 | 6
Completed | 8 | 3 | 3 | 3 | 3 | 6 | 5 | 9 | 6 | 6 | 4 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 1 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all enrolled participants who received at least one dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo IV SAD | PF-06835375 0.03 mg IV SAD | PF-06835375 0.1 mg IV SAD | PF-06835375 0.3 mg IV SAD | PF-06835375 1 mg IV SAD | PF-06835375 3 mg IV SAD | PF-06835375 6 mg IV SAD | Placebo SC MAD | PF-06835375 0.3 mg SC MAD | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD | Total
Number analyzed (Participants) | 8 | 3 | 3 | 3 | 3 | 6 | 5 | 11 | 6 | 6 | 7 | 6 | 6 | 73
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.00 (11.58) | 53.33 (11.02) | 47.33 (15.53) | 57.33 (6.03) | 54.00 (10.15) | 52.33 (13.95) | 54.00 (5.66) | 48.64 (13.60) | 52.00 (10.56) | 54.17 (7.70) | 53.57 (8.20) | 61.67 (10.80) | 58.50 (9.25) | 53.26 (10.71)
Age, Customized [Number; unit: Participants]
  <18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18-44 | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 4 | 2 | 0 | 1 | 1 | 1 | 15
  45-64 | 4 | 2 | 2 | 3 | 2 | 4 | 5 | 6 | 4 | 6 | 5 | 2 | 3 | 48
  >=65 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 2 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 3 | 2 | 3 | 6 | 5 | 11 | 5 | 4 | 7 | 5 | 4 | 65
  Male | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 10
  Not Hispanic or Latino | 7 | 3 | 3 | 3 | 3 | 3 | 5 | 9 | 5 | 5 | 5 | 6 | 6 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 15
  White | 4 | 2 | 2 | 1 | 2 | 4 | 4 | 9 | 6 | 4 | 6 | 5 | 5 | 54
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicity (DLT)
Description: DLT was defined as any of the following events meeting the criteria: (1) >=2 participants within a dose cohort developed Common Terminology Criteria for Adverse Events (CTCAE) v4.0 Grade 3 adverse event considered to be serious in the same organ system or 1 participant developed a CTCAE v4.0 Grade 4 or higher SAE considered related to study drug; (2) 50% or more participants within a dose cohort experienced a CTCAE v4.0 Grade 3 or higher infusion reaction; (3) a confirmed or probable case of Progressive Multifocal Leukoencephalopathy was observed; (4) the mean exposure for the treatment group reached or exceeded the exposure stopping limit of Cav of 261 mg/mL, or, based on the observed data, the group mean Cav of the next planned dose was projected to exceed the exposure stopping limit. Cav = average serum concentration.
Time Frame: From the first dose of study treatment up to 7-14 days after end of study criteria met (maximum duration for end of study criteria met: Day 225 for Part A, Day 281 for Part B)
Population: All participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV SAD | PF-06835375 0.03 mg IV SAD | PF-06835375 0.1 mg IV SAD | PF-06835375 0.3 mg IV SAD | PF-06835375 1 mg IV SAD | PF-06835375 3 mg IV SAD | PF-06835375 6 mg IV SAD | Placebo SC MAD | PF-06835375 0.3 mg SC MAD | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
Number analyzed (Participants) | 8 | 3 | 3 | 3 | 3 | 6 | 5 | 11 | 6 | 6 | 7 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) by Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Relatedness to study drug was assessed by the investigator. Treatment-emergent were events between first dose of study drug and up to approximately Week 40 that were absent before treatment or that worsened relative to pretreatment state. AEs are classified according to the severity in 3 categories a) mild - AEs does not interfere with participant's usual function b) moderate - AEs interferes to some extent with participant's usual function c) severe - AEs interferes significantly with participant's usual function.
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV SAD | PF-06835375 0.03 mg IV SAD | PF-06835375 0.1 mg IV SAD | PF-06835375 0.3 mg IV SAD | PF-06835375 1 mg IV SAD | PF-06835375 3 mg IV SAD | PF-06835375 6 mg IV SAD | Placebo SC MAD | PF-06835375 0.3 mg SC MAD | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
Number analyzed (Participants) | 8 | 3 | 3 | 3 | 3 | 6 | 5 | 11 | 6 | 6 | 7 | 6 | 6
Participants
  Mild (all causalities) | 3 | 0 | 1 | 0 | 0 | 3 | 0 | 4 | 2 | 1 | 1 | 1 | 3
  Moderate (all causalities) | 4 | 2 | 2 | 2 | 3 | 3 | 4 | 5 | 2 | 3 | 4 | 3 | 3
  Severe (all causalities) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Mild (treatment-related) | 2 | 0 | 1 | 0 | 0 | 4 | 1 | 3 | 3 | 0 | 2 | 1 | 1
  Moderate (treatment-related) | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 1 | 3 | 1 | 1
  Severe (treatment-related) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With All-Causality and Treatment-Related TEAEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Relatedness to study drug was assessed by the investigator. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to approximately Week 40 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV SAD | PF-06835375 0.03 mg IV SAD | PF-06835375 0.1 mg IV SAD | PF-06835375 0.3 mg IV SAD | PF-06835375 1 mg IV SAD | PF-06835375 3 mg IV SAD | PF-06835375 6 mg IV SAD | Placebo SC MAD | PF-06835375 0.3 mg SC MAD | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
Number analyzed (Participants) | 8 | 3 | 3 | 3 | 3 | 6 | 5 | 11 | 6 | 6 | 7 | 6 | 6
Participants
  Number of Participants with all-causality TEAEs | 8 | 3 | 3 | 2 | 3 | 6 | 5 | 9 | 4 | 4 | 5 | 4 | 6
  Number of Participants with all-causality SAEs | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Number of Participants with treatment-related TEAEs | 3 | 0 | 1 | 0 | 2 | 6 | 3 | 3 | 3 | 1 | 5 | 2 | 2
  Number of Participants with treatment-related SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Permanent Discontinuation Due to TEAEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent were events between first dose of study drug and up to approximately Week 40 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV SAD | PF-06835375 0.03 mg IV SAD | PF-06835375 0.1 mg IV SAD | PF-06835375 0.3 mg IV SAD | PF-06835375 1 mg IV SAD | PF-06835375 3 mg IV SAD | PF-06835375 6 mg IV SAD | Placebo SC MAD | PF-06835375 0.3 mg SC MAD | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
Number analyzed (Participants) | 8 | 3 | 3 | 3 | 3 | 6 | 5 | 11 | 6 | 6 | 7 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities in Hematology, Chemistry, and Urinalysis
Description: Hematology included hemoglobin, hematocrit, red blood cell, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet and white blood cell count, total neutrophils, eosinophils, monocytes, basophils and lymphocytes. Chemistry included blood urea nitrogen, creatinine, glucose, calcium, sodium, potassium, chloride, bicarbonate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid, albumin, total protein and creatine kinase. Urinalysis included pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, urobilinogen, urine bilirubin, microscopy and creatinine. Clinical significance was judged by the investigator and those met the criteria of AE are listed here. Clinically significant laboratory abnormalities reported for at least 1 participant in the whole study are presented here. Baseline was the last pre-dose measurement (first treatment for MAD cohorts).
Time Frame: From baseline up to end of study criteria met (maximum duration for end of study criteria met: Day 225 for Part A, Day 281 for Part B)
Population: All participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV SAD | PF-06835375 0.03 mg IV SAD | PF-06835375 0.1 mg IV SAD | PF-06835375 0.3 mg IV SAD | PF-06835375 1 mg IV SAD | PF-06835375 3 mg IV SAD | PF-06835375 6 mg IV SAD | Placebo SC MAD | PF-06835375 0.3 mg SC MAD | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
Number analyzed (Participants) | 8 | 3 | 3 | 3 | 3 | 6 | 5 | 11 | 6 | 6 | 7 | 6 | 6
Participants
  Elevated creatine phosphokinase (CPK) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Elevated liver enzymes (AST and ALT increased) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Elevated liver function tests (AST and ALT increased) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

6. Primary Outcome: Number of Participants With Post-Baseline Vital Signs Data Meeting Categorical Summarization Criteria
Description: Criteria for abnormality in vital signs: supine pulse rate <40 beats per minute (bpm) or >120 bpm; standing pulse rate <40 bpm or >120 bpm; sitting systolic blood pressure (BP) <90 mmHg, maximum increase or decrease from baseline of >=30 mmHg; sitting diastolic BP <50 mmHg, maximum increase or decrease from baseline of >=20 mmHg. Baseline was defined as the last pre-dose measurement in Day 1. Only those categories in which at least 1 participant had data were reported.
Time Frame: as for outcome 5
Population: All participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV SAD | PF-06835375 0.03 mg IV SAD | PF-06835375 0.1 mg IV SAD | PF-06835375 0.3 mg IV SAD | PF-06835375 1 mg IV SAD | PF-06835375 3 mg IV SAD | PF-06835375 6 mg IV SAD | Placebo SC MAD | PF-06835375 0.3 mg SC MAD | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
Number analyzed (Participants) | 8 | 3 | 3 | 3 | 3 | 6 | 5 | 11 | 6 | 6 | 7 | 6 | 6
Participants
  Sitting Systolic BP <90 mmHg | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Maximum Increase from Baseline in Sitting Systolic BP >= 30 mmHg | 4 | 1 | 1 | 1 | 2 | 3 | 1 | 1 | 2 | 2 | 3 | 0 | 1
  Maximum Decrease from Baseline in Sitting Systolic BP >= 30 mmHg | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 3 | 0 | 2 | 2 | 2 | 1
  Sitting Diastolic BP <50 mmHg | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Maximum Increase from Baseline in Sitting Diastolic BP >= 20 mmHg | 3 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 2 | 0 | 1 | 2
  Maximum Decrease from Baseline in Sitting Diastolic BP >= 20 mmHg | 2 | 0 | 0 | 2 | 2 | 4 | 2 | 4 | 1 | 1 | 2 | 2 | 2

7. Primary Outcome: Number of Participants With Post-Baseline Electrocardiogram (ECG) Data Meeting Categorical Summarization Criteria
Description: ECG abnormalities criteria included: 1) maximum QTc interval (ms): 450<= QTc <480, 480<= QTc <500, and QTc >=500; QTc maximum increase from baseline (ms): 30<= change <60, and change >=60; 2) maximum PR interval (ms): >=300; PR increase from baseline (ms): baseline >200 with 25% increase at maximum, baseline <=200 with 50% increase at maximum; 3) maximum QRS (ms): >=140; QRS increase from baseline (ms) >=50%. QTcF indicates QT interval corrected using the Fridericia's formula. QTcB indicates QT interval corrected using the Bazett's formula. Baseline was defined as the average of the triplicate pre-dose recordings at Day 1. Only those categories in which at least 1 participant had data were reported.
Time Frame: as for outcome 5
Population: All participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV SAD | PF-06835375 0.03 mg IV SAD | PF-06835375 0.1 mg IV SAD | PF-06835375 0.3 mg IV SAD | PF-06835375 1 mg IV SAD | PF-06835375 3 mg IV SAD | PF-06835375 6 mg IV SAD | Placebo SC MAD | PF-06835375 0.3 mg SC MAD | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
Number analyzed (Participants) | 8 | 3 | 3 | 3 | 3 | 6 | 5 | 11 | 6 | 6 | 7 | 6 | 6
Participants
  Maximum QRS (ms) >=140 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  450<= Maximum QTcB Interval (ms) <480 | 4 | 1 | 2 | 0 | 2 | 1 | 3 | 6 | 1 | 1 | 3 | 2 | 3
  480<= Maximum QTcB Interval (ms) <500 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0
  Maximum QTcB Interval (ms) >=500 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  30<= QTcB Maximum Increase From Baseline (ms) <60 | 4 | 0 | 0 | 0 | 0 | 2 | 4 | 3 | 2 | 1 | 0 | 2 | 3
  450<= Maximum QTcF Interval (ms) <480 | 2 | 2 | 1 | 1 | 1 | 0 | 1 | 4 | 0 | 0 | 3 | 0 | 0
  30<= QTcF Maximum Increase From Baseline (ms) <60 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  480<= Maximum QTcF Interval (ms) <500 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0

8. Primary Outcome: Number of Participants With All-Causality and Treatment-Related Infections and Infestations
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Relatedness to study drug was assessed by the investigator. The incidence of AEs by system organ class "infections and infestations" was reported here.
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo IV SAD | PF-06835375 0.03 mg IV SAD | PF-06835375 0.1 mg IV SAD | PF-06835375 0.3 mg IV SAD | PF-06835375 1 mg IV SAD | PF-06835375 3 mg IV SAD | PF-06835375 6 mg IV SAD | Placebo SC MAD | PF-06835375 0.3 mg SC MAD | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
Number analyzed (Participants) | 8 | 3 | 3 | 3 | 3 | 6 | 5 | 11 | 6 | 6 | 7 | 6 | 6
Participants
  Number of Participants with all-causality Infections and Infestations | 4 | 2 | 3 | 0 | 2 | 1 | 3 | 3 | 2 | 3 | 2 | 0 | 2
  Number of Participants with treatment-related Infections and Infestations | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: B Cell Maximum Decrease (%) From Baseline Over Time Following Single and Multiple Doses of PF-06835375
Description: Blood samples for the assessment of B cell were collected and analyzed by flow cytometry. Baseline was defined as the average of screening and pre-dose measures.
Time Frame: Screening, Day 1, 2, 4, 8, 15, 29, 36 (Part B only), 43, 57, 85, 113, and every 4 weeks until criteria for end of study met (maximum duration for end of study criteria met: Day 225 for Part A, Day 281 for Part B)
Population: All enrolled participants who received at least 1 dose of study treatment and had at least 1 pharmacodynamic measurement.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of decrease from baseline
Arm/Group | Placebo IV SAD | PF-06835375 0.03 mg IV SAD | PF-06835375 0.1 mg IV SAD | PF-06835375 0.3 mg IV SAD | PF-06835375 1 mg IV SAD | PF-06835375 3 mg IV SAD | PF-06835375 6 mg IV SAD | Placebo SC MAD | PF-06835375 0.3 mg SC MAD | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
Number analyzed (Participants) | 8 | 3 | 3 | 3 | 3 | 6 | 5 | 11 | 6 | 6 | 7 | 6 | 6
Percentage of decrease from baseline | 37.693 (43.0477) | 67.283 (29.3555) | 84.978 (5.9053) | 94.052 (2.4246) | 98.546 (0.1627) | 98.588 (1.0295) | 99.326 (0.3272) | 41.854 (52.5341) | 91.056 (12.6425) | 99.650 (0.4036) | 99.287 (0.6300) | 99.278 (1.4476) | 99.134 (0.9983)

10. Secondary Outcome: cTfh Cell Depletion Maximum Decrease (%) From Baseline Over Time Following Single and Multiple Doses of PF-06835375
Description: Blood samples for the assessment of circulating follicular T helper like (cTfh) cell were collected and analyzed by flow cytometry. Baseline was defined as the average of screening and pre-dose measures.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of decrease from baseline
Arm/Group | Placebo IV SAD | PF-06835375 0.03 mg IV SAD | PF-06835375 0.1 mg IV SAD | PF-06835375 0.3 mg IV SAD | PF-06835375 1 mg IV SAD | PF-06835375 3 mg IV SAD | PF-06835375 6 mg IV SAD | Placebo SC MAD | PF-06835375 0.3 mg SC MAD | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
Number analyzed (Participants) | 8 | 3 | 3 | 3 | 3 | 6 | 5 | 11 | 6 | 6 | 7 | 6 | 6
Percentage of decrease from baseline | 45.227 (48.6385) | 62.360 (23.1206) | 84.994 (11.2007) | 89.324 (6.3399) | 98.675 (1.2762) | 97.283 (3.0481) | 97.789 (3.1257) | 58.116 (52.5069) | 89.540 (14.8599) | 95.442 (5.3905) | 96.683 (1.8503) | 97.721 (1.6523) | 98.118 (0.8825)

11. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of PF-06835375 in Part A (SAD)
Description: Cmax is maximum observed serum concentration. Cmax for PF-06835375 was observed directly from data.
Time Frame: Day 1 (pre-dose, 2, 4, 6, 8, 12 hours post dose), 2, 4, 8, 15, 29, 43, 57, 85, 113 and 141 for Day 1 PK estimates
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | PF-06835375 0.03 mg IV SAD | PF-06835375 0.1 mg IV SAD | PF-06835375 0.3 mg IV SAD | PF-06835375 1 mg IV SAD | PF-06835375 3 mg IV SAD | PF-06835375 6 mg IV SAD
Number analyzed (Participants) | 2 | 1 | 3 | 3 | 6 | 4
nanogram/milliliter (ng/mL) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 103.0 (197) | 208.7 (28) | 994.7 (29) | 2645 (13)

12. Secondary Outcome: Time to Reach Cmax (Tmax) of PF-06835375 in Part A (SAD)
Description: Tmax is the time for Cmax. Tmax for PF-06835375 was observed directly from data as time of first occurrence.
Time Frame: Day 1 (pre-dose, 2, 4, 6, 8, 12 hours post dose), 2, 4, 8, 15, 29, 43, 57, 85, 113 and 141 for Day 1 PK estimates
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest.
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | PF-06835375 0.03 mg IV SAD | PF-06835375 0.1 mg IV SAD | PF-06835375 0.3 mg IV SAD | PF-06835375 1 mg IV SAD | PF-06835375 3 mg IV SAD | PF-06835375 6 mg IV SAD
Number analyzed (Participants) | 2 | 1 | 3 | 3 | 6 | 4
hour (hr) | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA [NA to NA] — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 2.17 [2.15 to 2.20] | 2.08 [2.07 to 4.15] | 2.24 [2.17 to 4.12] | 3.96 [2.00 to 8.12]

13. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of PF-06835375 in Part A (SAD)
Description: AUCinf is the area under the serum concentration-time profile from time zero extrapolated to infinite time.
Time Frame: Day 1 (pre-dose, 2, 4, 6, 8, 12 hours post dose), 2, 4, 8, 15, 29, 43, 57, 85, 113 and 141 for Day 1 PK estimates
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | PF-06835375 0.03 mg IV SAD | PF-06835375 0.1 mg IV SAD | PF-06835375 0.3 mg IV SAD | PF-06835375 1 mg IV SAD | PF-06835375 3 mg IV SAD | PF-06835375 6 mg IV SAD
Number analyzed (Participants) | 2 | 0 | 3 | 3 | 6 | 4
nanogram*hour/milliliter (ng*hr/mL) | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. |  | 1573 (2409) | 7467 (84) | 88190 (35) | 288000 (30)

14. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-06835375 in Part A (SAD)
Description: AUClast is the area under the curve from time zero to last quantifiable concentration. AUClast for PF-06835375 was determined using linear/log trapezoidal method.
Time Frame: Day 1 (pre-dose, 2, 4, 6, 8, 12 hours post dose), 2, 4, 8, 15, 29, 43, 57, 85, 113 and 141 for Day 1 PK estimates
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06835375 0.03 mg IV SAD | PF-06835375 0.1 mg IV SAD | PF-06835375 0.3 mg IV SAD | PF-06835375 1 mg IV SAD | PF-06835375 3 mg IV SAD | PF-06835375 6 mg IV SAD
Number analyzed (Participants) | 2 | 1 | 3 | 3 | 6 | 4
ng*hr/mL | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 1380 (2950) | 7327 (85) | 87120 (36) | 287400 (30)

15. Secondary Outcome: Cmax of PF-06835375 Following First Dose and Multiple Doses in Part B (MAD)
Description: Cmax is maximum observed serum concentration. Cmax for PF-06835375 was observed directly from data. There were less than 3 quantifiable concentrations for participants in PF-06835375 0.3 mg SC MAD cohort, therefore the serum PK parameters were not calculated.
Time Frame: Day 1 (pre-dose, 2, 4, 6, 8, 12 hours post dose), 2, 4, 8 and 15 for Day 1 PK estimates; Day 29 (pre-dose, 2, 4, 6, 8, hours post dose), 36, 43, 57, 85 and 113 for Day 29 PK estimates
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
Number analyzed (Participants) | 4 | 7 | 6 | 5
ng/mL
  Day 1 | 5.743 (148) | 34.82 (79) | 77.72 (150) | 257.8 (204)
  Day 29: number analyzed (Participants) | 3 | 7 | 6 | 5
  Day 29 | 26.92 (68) | 89.68 (93) | 209.6 (115) | 262.1 (224)

16. Secondary Outcome: Tmax of PF-06835375 Following First Dose and Multiple Doses in Part B (MAD)
Description: Tmax is the time for Cmax. Tmax for PF-06835375 was observed directly from data as time of first occurrence. There were less than 3 quantifiable concentrations for participants in PF-06835375 0.3 mg SC MAD cohort, therefore the serum PK parameters were not calculated.
Time Frame: as for outcome 15
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest.
Measure: Median (Full Range); unit: hr
Arm/Group | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
Number analyzed (Participants) | 4 | 7 | 6 | 5
hr
  Day 1 | 170 [67.4 to 170] | 168 [72.7 to 361] | 169 [73.3 to 192] | 144 [47.7 to 172]
  Day 29: number analyzed (Participants) | 3 | 7 | 6 | 5
  Day 29 | 169 [168 to 169] | 169 [123 to 337] | 171 [120 to 336] | 121 [7.55 to 169]

17. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) of PF-06835375 Following First Dose and Multiple Doses in Part B (MAD)
Description: AUCtau is area under the serum concentration-time profile from time 0 to time tau, the dosing interval, where tau= 28 days. AUCtau for PF-06835375 was determined using linear/log trapezoidal method. There were less than 3 quantifiable concentrations for participants in PF-06835375 0.3 mg SC MAD cohort, therefore the serum PK parameters were not calculated.
Time Frame: as for outcome 15
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
Number analyzed (Participants) | 4 | 7 | 6 | 5
ng*hr/mL
  Day 1: number analyzed (Participants) | 4 | 7 | 5 | 5
  Day 1 | 1964 (130) | 11010 (84) | 28070 (251) | 70630 (202)
  Day 29: number analyzed (Participants) | 3 | 6 | 6 | 5
  Day 29 | 9309 (62) | 25610 (125) | 76450 (142) | 88540 (154)

18. Secondary Outcome: AUClast of PF-06835375 Following Multiple Doses in Part B (MAD)
Description: AUClast is the area under the curve from time zero to last quantifiable concentration. AUClast for PF-06835375 was determined using linear/log trapezoidal method. There were less than 3 quantifiable concentrations for participants in PF-06835375 0.3 mg SC MAD cohort, therefore the serum PK parameters were not calculated.
Time Frame: Day 29 (pre-dose, 2, 4, 6, 8, hours post dose), 36, 43, 57, 85 and 113 for Day 29 PK estimates
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
Number analyzed (Participants) | 3 | 7 | 6 | 5
ng*hr/mL | 9346 (61) | 22050 (146) | 84370 (160) | 96610 (141)

19. Secondary Outcome: Minimum Observed Serum Trough Concentration (Cmin) of PF-06835375 Following Multiple Doses in Part B (MAD)
Description: Cmin is minimum observed serum trough concentration. Cmin was observed directly from data. There were less than 3 quantifiable concentrations for participants in PF-06835375 0.3 mg SC MAD cohort, therefore the serum PK parameters were not calculated.
Time Frame: Day 29 (pre-dose, 2, 4, 6, 8, hours post dose), 36, 43, 57, 85 and 113 for Day 29 PK estimates
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
Number analyzed (Participants) | 2 | 5 | 6 | 5
ng/mL | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated | 6.075 (80) | 11.81 (434) | 9.410 (199)

20. Secondary Outcome: Observed Accumulation Ratio (Rac) of PF-06835375 Following Multiple Doses in Part B (MAD)
Description: Rac is observed accumulation ratio. Rac = Day 29 AUCtau / Day 1 AUCtau. There were less than 3 quantifiable concentrations for participants in PF-06835375 0.3 mg SC MAD cohort, therefore the serum PK parameters were not calculated.
Time Frame: as for outcome 15
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
Number analyzed (Participants) | 2 | 6 | 5 | 4
ratio | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 2.410 (74) | 2.977 (79) | 2.001 (209)

21. Secondary Outcome: Peak-to-trough Fluctuation (PTF) of PF-06835375 Following Multiple Doses in Part B (MAD)
Description: PTF is peak-to-trough fluctuation at steady state. PTF = (Cmax-Cmin)/Cav. Cav is average serum concentration. There were less than 3 quantifiable concentrations for participants in PF-06835375 0.3 mg SC MAD cohort, therefore the serum PK parameters were not calculated.
Time Frame: Day 29 (pre-dose, 2, 4, 6, 8, hours post dose), 36, 43, 57, 85 and 113 for Day 29 PK estimates
Population: All enrolled participants treated who had at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
Number analyzed (Participants) | 2 | 5 | 6 | 5
ratio | NA (NA) — NA indicates not calculable. There were insufficient number of participants with reportable parameter values (less than 3), so these summary statistics were not calculated. | 2.037 (26) | 1.687 (31) | 1.830 (35)

22. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) and Neutralizing Antibody (NAb) Against PF-06835375
Description: To evaluate the immunogenicity as measured by presence of ADA and NAb in participants treated with PF-06835375.
Time Frame: Day 1, 15, 29, 43, 57, 85, 113, and every 4 weeks until criteria for end of study met (maximum duration for end of study criteria met: Day 225 for Part A, Day 281 for Part B)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06835375 0.03 mg IV SAD | PF-06835375 0.1 mg IV SAD | PF-06835375 0.3 mg IV SAD | PF-06835375 1 mg IV SAD | PF-06835375 3 mg IV SAD | PF-06835375 6 mg IV SAD | PF-06835375 0.3 mg SC MAD | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 5 | 6 | 6 | 7 | 6 | 6
Participants
  Number of ADA or NAb evaluable participants with positive ADA | 0 | 0 | 1 | 1 | 3 | 2 | 3 | 3 | 1 | 1 | 2
  Number of ADA or NAb evaluable participants with positive NAb | 0 | 0 | 1 | 1 | 3 | 2 | 2 | 1 | 1 | 1 | 2

ADVERSE EVENTS:
Time Frame: From the first dose of study treatment up to 7-14 days after end of study criteria met (maximum duration for end of study criteria met: Day 225 for Part A, Day 281 for Part B)
Arm/Group | Placebo IV SAD | PF-06835375 0.03 mg IV SAD | PF-06835375 0.1 mg IV SAD | PF-06835375 0.3 mg IV SAD | PF-06835375 1 mg IV SAD | PF-06835375 3 mg IV SAD | PF-06835375 6 mg IV SAD | Placebo SC MAD | PF-06835375 0.3 mg SC MAD | PF-06835375 1 mg SC MAD | PF-06835375 3 mg SC MAD | PF-06835375 6 mg SC MAD | PF-06835375 10 mg SC MAD
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/3 | 0/3 | 0/3 | 0/3 | 0/6 | 0/5 | 0/11 | 0/6 | 0/6 | 0/7 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/8 | 1/3 | 0/3 | 1/3 | 0/3 | 0/6 | 0/5 | 0/11 | 0/6 | 0/6 | 0/7 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 8/8 | 3/3 | 3/3 | 2/3 | 3/3 | 6/6 | 5/5 | 9/11 | 4/6 | 4/6 | 5/7 | 4/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo IV SAD (N=8) | PF-06835375 0.03 mg IV SAD (N=3) | PF-06835375 0.1 mg IV SAD (N=3) | PF-06835375 0.3 mg IV SAD (N=3) | PF-06835375 1 mg IV SAD (N=3) | PF-06835375 3 mg IV SAD (N=6) | PF-06835375 6 mg IV SAD (N=5) | Placebo SC MAD (N=11) | PF-06835375 0.3 mg SC MAD (N=6) | PF-06835375 1 mg SC MAD (N=6) | PF-06835375 3 mg SC MAD (N=7) | PF-06835375 6 mg SC MAD (N=6) | PF-06835375 10 mg SC MAD (N=6)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo IV SAD (N=8) | PF-06835375 0.03 mg IV SAD (N=3) | PF-06835375 0.1 mg IV SAD (N=3) | PF-06835375 0.3 mg IV SAD (N=3) | PF-06835375 1 mg IV SAD (N=3) | PF-06835375 3 mg IV SAD (N=6) | PF-06835375 6 mg IV SAD (N=5) | Placebo SC MAD (N=11) | PF-06835375 0.3 mg SC MAD (N=6) | PF-06835375 1 mg SC MAD (N=6) | PF-06835375 3 mg SC MAD (N=7) | PF-06835375 6 mg SC MAD (N=6) | PF-06835375 10 mg SC MAD (N=6)
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Injection site scab (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 1 | 1 | 3 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Electrocardiogram T wave amplitude decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 4 | 2 | 2 | 2 | 1 | 1 | 1 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mass (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tenderness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaccination site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 1 | 0 | 0
Vaccination site induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaccination site nodule (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaccination site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Vaccination site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaccination site warmth (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gallbladder disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Allergy to vaccine (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Bacterial vulvovaginitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device malfunction (Product Issues) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalciuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stag horn calculus (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/51/NCT03334851/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/51/NCT03334851/SAP_001.pdf